CLINICAL TRIAL: NCT00328744
Title: Reducing Snack Food Variety During Obesity Treatment
Brief Title: Reducing Snack Variety in Weight Loss Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK074721-01 (NIH)
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2008-10

CONDITIONS: Obesity
Keywords: Weight; Dietary intake; Energy; Hedonics; Behavioral; Sensory-specific satiety; Monotony
MeSH Terms: conditions — Obesity; Body Weight; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): Behavioral: Behavioral weight loss (Standard)
  Interventions: Behavioral: Standard
- 2 (Experimental): Behavioral: Behavioral weight loss (Limited Variety)
  Interventions: Behavioral: Standard; Behavioral: Limited Variety

INTERVENTIONS:
Behavioral: Standard — 18-month standard behavioral weight loss intervention
Behavioral: Limited Variety — Two chosen snack foods
  Arms: 2

SUMMARY:
The rising prevalence of obesity in the United States is believed to be due to increased exposure to adverse environmental factors, such as food portion sizes and increased dietary variety. Although decreasing portion sizes is a strategy used in weight loss programs, research has not studied the effects of decreasing dietary variety. Cross-sectional studies show a positive association between variety and body weight and in our own studies the investigators have shown that greater reductions in the number of different snack foods (i.e., cookies, chips) consumed predicted greater decreases in overall caloric and fat intake and greater weight loss. Limiting variety may reduce intake through long-term sensory-specific satiety and/or monotony. Reducing dietary variety is a novel dietary approach with the potential to improve long-term weight loss, which has not been studied as a clinical strategy in obesity research. The objective of this application is to conduct a randomized controlled trial of a behavioral weight loss intervention limiting the number of different snack foods consumed. Two hundred overweight and obese participants will be randomized to a standard behavioral intervention (Standard) or to a standard behavioral intervention that also limits the number of different snack foods consumed (Limited Variety). Both conditions will receive an 18-month standard behavioral intervention, using behavioral techniques (i.e., self-monitoring) to change eating behaviors. Participants in the Limited Variety condition will also limit variety in snack foods to only two chosen snack foods throughout the intervention. Measures of weight, snack food consumption and hedonics, and diet satisfaction will be taken at 0, 6, 12, and 18 months. This investigation will determine:

1. if the Limited Variety condition produces greater weight loss than the Standard condition at 18 months;
2. if the Limited Variety condition consumes fewer servings and calories from snack foods than the Standard condition;
3. if limiting snack food variety produces long-term sensory-specific satiety and/or monotony.

Relevance: Experimental studies show that limiting dietary variety profoundly reduces intake. To date, there is no dietary prescription that has been tested that capitalizes on the effect of variety on intake that can be maintained. This will be the first investigation to examine methods of manipulating dietary variety that can be adhered to over time and that influence intake, weight loss, and weight loss maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21 and 65 years. Older adults may have more medical co-morbidities, requiring greater medical supervision. Although pediatric obesity is a significant concern, this group has different nutritional needs and requires different levels of therapist and parental involvement than are proposed.
2. Body mass index (BMI) between 27 and 45 kg/m2. Based upon the Evidence Report (72), weight loss is recommended for individuals with a BMI > 25. A BMI of > 27 was chosen as eligibility criteria for this investigation because this level of BMI will allow for a 10% weight loss to occur prior to reaching a BMI of < 25. Individuals with a BMI of > 45 have more medical co-morbidities and require greater medical supervision, and thus will be considered ineligible for this investigation.

Exclusion Criteria:

1. Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q) (73). Individuals endorsing joint problems, prescription medication usage, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.
2. Have an allergy to a food commonly found in snack foods (i.e., nuts, milk and egg proteins).
3. Report major psychiatric diseases or organic brain syndromes.
4. Are currently participating in a weight loss program and/or taking weight loss medication or lost > 5% of body weight during the past 6 months.
5. Intend to move outside of the metropolitan area within the time frame of the investigation.
6. Are pregnant, lactating, less than 6 months post-partum, or plan to become pregnant during the time frame of the investigation.
7. Consume < 5 different types of snack food per week. Pilot data indicated that upon screening 44 participants, mean weekly variety of snack foods was 8.7 (range 2 to 14, with only two participants consuming < 5 snack foods per week).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2006-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Weight loss | 18 months

SECONDARY OUTCOMES:
Diet | 18 months
Hedonics of food | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, PhD, Principal Investigator — University of Tennessee
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Raynor HA, Van Walleghen EL, Bachman JL, Looney SM, Phelan S, Wing RR. Dietary energy density and successful weight loss maintenance. Eat Behav. 2011 Apr;12(2):119-25. doi: 10.1016/j.eatbeh.2011.01.008. Epub 2011 Jan 25. PMID 21385641